CLINICAL TRIAL: NCT02505711
Title: Reducing Young Child Undernutrition Through an Integrated Agricultural Project With Women's Groups: A Cluster-randomized Trial in Rural Bangladesh
Brief Title: Food and Agricultural Approaches to Reducing Malnutrition
Acronym: FAARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sabine Gabrysch (Other)
Collaborators: Helen Keller International (Other); BRAC University (Other); University of Giessen (Other); German Federal Ministry of Education and Research (Other Government); Department for International Development, United Kingdom (Other Government); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); German Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Sabine Gabrysch, Head, Unit of Epidemiology and Biostatistics, Institute of Global Health, Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01ER1201
Record Dates: First submitted 2015-07-17; First posted 2015-07-22 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Malnutrition
Keywords: Agriculture; Food; Micronutrients; Pregnancy; Infants; Women's groups; Bangladesh
MeSH Terms: conditions — Malnutrition | interventions — Agriculture; Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homestead Food Production (Experimental): Enrolled in Homestead Food Production program from 2015 to 2019, 48 clusters, approx. 1350 women and 750 children
  Interventions: Behavioral: Homestead Food Production program
- Control (No Intervention): (Health system strengthening in the study area), 48 clusters, approx. 1350 women and 750 children

INTERVENTIONS:
Behavioral: Homestead Food Production program — Training and support for vegetable gardening and poultry rearing, and education on young child nutrition, hygiene and health topics, in women's groups, as designed by the international non-governmental organization (NGO) Helen Keller International (HKI).
  Other Names: Agriculture; Home gardening; Nutrition education
  Arms: Homestead Food Production

SUMMARY:
The aim of this study is to evaluate the potential of reducing young child undernutrition in low-income countries through an integrated program that trains women's groups in agriculture, nutrition, child care and hygiene.

DETAILED DESCRIPTION:
An estimated 165 million children worldwide suffer from chronic undernutrition which leads to compromised physical and cognitive development and prevents them from reaching their full potential. Nutrition-sensitive agricultural interventions that aim to increase dietary diversity, empower women and include an educational behaviour change component focused on nutrition and hygiene are a promising and sustainable approach to addressing undernutrition. However, evidence on the impact of such interventions is still scarce due to a lack of rigorous long-term evaluations.

This study will test the hypothesis that integrated agriculture, nutrition and hygiene interventions can reduce undernutrition when children benefit in their crucial first 1000 days. The investigators will conduct an impact evaluation of Helen Keller International's Homestead Food Production program in Bangladesh that trains women's groups in vegetable and fruit gardening, poultry rearing, hygiene, child care and nutrition. Furthermore, the investigators will assess the program impact pathway to discern how any impact is achieved (through improved food production, income, food security, health service use, female empowerment, feeding and hygiene practices).

The study design is a cluster-randomized controlled field trial in two sub-districts of Habiganj District, Sylhet Division, Bangladesh, including 2700 young women in 96 settlements. After the baseline survey in 2015, settlements will be randomized into 48 intervention and 48 control settlements. Women in the intervention settlements will receive training and support in Homestead Food Production during the following four years. A surveillance system will collect data on pregnancies, births, child development, nutrition and infections as well as pathway indicators. In 2019, the investigators will conduct the endline survey to assess the nutritional status of the 2700 women and their then approximately 1500 children below 3 years of age and compare between intervention and control.

ELIGIBILITY:
Inclusion Criteria:

For settlements:

* Located in selected unions of Habiganj District, Sylhet Division, North East Bangladesh
* Minimum distance to adjacent settlement at least 400 m
* Judged to be suitable for Homestead Food Production program by the NGO HKI Bangladesh (dry land year-round, at least 10 women eligible and interested)

For women:

* Married and aged 30 years or less at enumeration
* Woman's husband stays overnight in household at least once a year
* Access to at least 1 decimal of land, ideally 0.25 decimal near the house

For children:

* Biological child of a participant woman
* Aged 0-35 months at survey start or surveillance visit

Exclusion Criteria:

For women:

* Lack of interest in participating in a gardening program

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2705 (Actual)
Dates: Start 2015-03-14 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Linear growth in children below 3 years of age | Measured 50 months after randomization (endline survey 2019)
  Length/height-for-age Z-score

SECONDARY OUTCOMES:
Linear growth in children aged 6-30 months | Measured 50 months after randomization
  Length/height-for-age Z-score
Intrauterine growth retardation: length | Measured within 3 days of birth, 15-57 months after randomization
  Length-for-gestational-age
Intrauterine growth retardation: small-for-gestational age | Measured within 3 days of birth, 15-57 months after randomization
  Weight-for-gestational-age adjusted for time since birth
Intrauterine growth retardation: head size | Measured within 3 days of birth, 15-57 months after randomization
  Head circumference-for-gestational-age
Wasting in children below 3 years of age | Measured 50 months after randomization
  Weight-for-length/height Z-score
Head circumference in children below 3 years of age | Measured 50 months after randomization
  Head circumference-for-age Z-score
Underweight in women | Measured 50 months after randomization
  Body Mass Index (BMI, non-pregnant women), mid-upper-arm circumference (MUAC, pregnant women)
Gestational weight gain | Measured every 2 months during pregnancy, 6-57 months after randomization
  Gestational weight gain Z-score
Anemia in women and children below 3 years of age | Measured 50 months after randomization
  Hemoglobin concentration
Micronutrients: Vitamin A deficiency in women and in children below 3 years of age | Measured 50 months after randomization
  Retinol-binding protein, corrected for inflammation (CRP, AGP)
Micronutrients: Iron deficiency in women and in children below 3 years of age | Measured 50 months after randomization
  Ferritin and soluble transferrin receptor, corrected for inflammation (CRP, AGP)
Micronutrients: Zinc deficiency in women and in children below 3 years of age | Measured 50 months after randomization
  Serum zinc, corrected for inflammation (CRP, AGP)
Early child development (adapted WHO milestones) | Measured at appropriate ages for milestones, 6-50 months after randomization
  Gross and fine motor, cognitive, personal-social and communication skills
Diarrhea in children below 3 years of age | Measured every 2 months, 6-50 months after randomization
  Period and point prevalence of diarrhea
Acute respiratory infection in children below 3 years of age | Measured every 2 months, 6-50 months after randomization
  Period prevalence of acute respiratory infection
Enteropathy in children below 18 months of age | Measured 36 and 50 months after randomization
  Biomarkers: faecal myeloperoxidase, faecal α1-antitrypsin, faecal neopterin, serum C-reactive protein, serum α-1-acid glycoprotein
Dietary adequacy in women and children below 3 years of age | Measured every 2 months, 6-50 months after randomization
  Mean probability of adequate micronutrient intake (MPA)
Dietary diversity in women and children below 3 years of age | Measured every 2 months, 6-50 months after randomization
  Individual dietary diversity score, breastfeeding behaviors
Fecal contamination of complementary food for children 6-18 months of age | Measured 36 months after randomization
  Log-transformed counts of total coliforms and E. coli in complementary food samples
Food hygiene behaviour in mothers of children aged 6-18 months | Measured 36 months after randomization
  Hygiene score from structured observation of mothers

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Gabrysch, MD MSc PhD, Principal Investigator — Heidelberg University

REFERENCES:
- [Derived] Wendt AS, Waid JL, Muller-Hauser AA, Lambrecht NJ, Huda TMN, Kyei NNA, Gabrysch S. Impacts of a Homestead Food Production Intervention on Anaemia and Micronutrient Deficiencies Among Women and Children in Rural Bangladesh: A Cluster-Randomized Controlled Trial. Matern Child Nutr. 2025 Oct;21(4):e70043. doi: 10.1111/mcn.70043. Epub 2025 May 19. PMID 40387380
- [Derived] Sobhan S, Muller-Hauser AA, Gon G, Nurul Huda TM, Waid JL, Wendt AS, Rahman M, Gabrysch S. Effect of a behaviour change intervention on household food hygiene practices in rural Bangladesh: A cluster-randomised controlled trial. Int J Hyg Environ Health. 2024 Jan;255:114291. doi: 10.1016/j.ijheh.2023.114291. Epub 2023 Nov 18. PMID 37983985
- [Derived] Waid JL, Wendt AS, Kader A, Sobhan S, Gabrysch S. Impact of a Homestead Food Production Program on Dietary Diversity: Seasonal and Annual Results from the Cluster-Randomized FAARM Trial in Sylhet, Bangladesh. J Nutr. 2024 Jan;154(1):191-201. doi: 10.1016/j.tjnut.2023.10.014. Epub 2023 Oct 21. PMID 37871747
- [Derived] Muller-Hauser AA, Huda TMN, Sobhan S, Lambrecht NJ, Waid JL, Wendt AS, Ali S, Rahman M, Gabrysch S. Effect of a Homestead Food Production and Food Hygiene Intervention on Biomarkers of Environmental Enteric Dysfunction in Children Younger Than 24 Months in Rural Bangladesh: A Cluster-Randomized Controlled Trial. Am J Trop Med Hyg. 2023 Oct 2;109(5):1166-1176. doi: 10.4269/ajtmh.23-0153. Print 2023 Nov 1. PMID 37783459
- [Derived] Lambrecht NJ, Muller-Hauser AA, Sobhan S, Schmidt WP, Huda TMN, Waid JL, Wendt AS, Kader A, Gabrysch S. Effect of a Homestead Food Production Program on the Prevalence of Diarrhea and Acute Respiratory Infection in Children in Sylhet, Bangladesh: A Cluster-Randomized Controlled Trial. Am J Trop Med Hyg. 2023 Aug 14;109(4):945-956. doi: 10.4269/ajtmh.23-0152. Print 2023 Oct 4. PMID 37580032
- [Derived] Dupuis S, Hennink M, Wendt AS, Waid JL, Kalam MA, Gabrysch S, Sinharoy SS. Women's empowerment through homestead food production in rural Bangladesh. BMC Public Health. 2022 Jan 19;22(1):134. doi: 10.1186/s12889-022-12524-2. PMID 35045859
- [Derived] Wendt AS, Waid JL, Gabrysch S. Dietary Factors Moderate the Relation between Groundwater Iron and Anemia in Women and Children in Rural Bangladesh. Curr Dev Nutr. 2019 Aug 6;3(10):nzz093. doi: 10.1093/cdn/nzz093. eCollection 2019 Oct. PMID 31620671
- [Derived] Wendt AS, Sparling TM, Waid JL, Mueller AA, Gabrysch S. Food and Agricultural Approaches to Reducing Malnutrition (FAARM): protocol for a cluster-randomised controlled trial to evaluate the impact of a Homestead Food Production programme on undernutrition in rural Bangladesh. BMJ Open. 2019 Jul 4;9(7):e031037. doi: 10.1136/bmjopen-2019-031037. PMID 31278109